CLINICAL TRIAL: NCT07121348
Title: Effect of Different NanoScaffolds on Pulp Regeneration in Non-Vital Immature Permanent Teeth (Randomized Clinical Trial)
Acronym: Regeneration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nada Ahmed Hashad, Effect of Different NanoScaffolds on Pulp Regeneration in Non-Vital Immature Permanent Teeth (Randomized Clinical Trial), Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REGEN2025-NH
Record Dates: First submitted 2025-08-04; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Necrotic Immature Permanent Incisors
MeSH Terms: interventions — Nanoparticles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Platelet Rich Fibrin (PRF only) (Experimental): patients will recieve canal disinfection followed by induction of bleeding and placement of platelet rich fibrin as the only scaffold before coronal sealing.
  platelet rich fibrin is obtained br removing the middle layer from a centrifuged blood sample and this is rich in platelets that play role in promoting tissue regeneration.
  Interventions: Procedure: Platelet rich fibrin
- Mesoporous Silica Nanoparticles scaffold (MSN) (Experimental): patients will recieve canal disinfection followed by induction of bleeding and injection of this scaffold directly before coronal sealing.
  Mesoporous Silica Nanoparticles are biocompatible with high surface area that used as scaffold for enhancing the outcome.
  Interventions: Procedure: Platelet rich fibrin
- Hyaluronic Acid Nanoparticles scaffold (HA) (Experimental): patients will recieve canal disinfection followed by induction of bleeding and injection of this scaffold directly before coronal sealing.
  Hyalornic Acid nanoparticles are biodegradable with high water retention capacity promoting pulp tissue regeneration.
  Interventions: Procedure: Platelet rich fibrin
- Pomegranate ( punica granatum) Extract Nanoparticles scaffold (Experimental): patients will recieve canal disinfection followed by induction of bleeding and injection of this scaffold directly before coronal sealing.
  Pomegranate Extract Nanoparticles are synthesized from Punica granatum exract with potential antimicrobial and regenerative properties.
  Interventions: Procedure: Platelet rich fibrin

INTERVENTIONS:
Procedure: Platelet rich fibrin — platelet rich fibrin is obtained by removing the middle layer from a centrifuged blood sample and is rich with platelets that plays an important role in tissue regeneration mesoporous silica nanoparticles are high surface area and excellent biocompatibility and enhance the outcome hyalurnic acid nanoparticles are high water capacity and involved in cell proliferation and adhesion and help in tissue regeneration pomegranate nanoparticles has anti-inflammatory and antibacterial effect and also help in tissue proliferation and regeneration
  Other Names: mesoporous silica nanoparticles; hyaluronic acid nanoparticles; pomegranate (punica granatum) nanoparticles

SUMMARY:
the clinical trial aims to evaluate efficency of different scaffolds in cases of regeneration

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical and radiographic outcome of regenerative endodontic procedures in immature non-vital permanent teeth using different nanoscaffolds (Platelet-rich fibrin, Mesoporous silica nanoparticles, Hyaluronic acid nanoparticles, Pomegranate nanoparticles)

ELIGIBILITY:
Inclusion Criteria:• Patients free from any systemic diseases that may interfer with the normal healing process.

* Maxillary traumatized or cariously exposed non-vital immature anterior teeth.
* Teeth don't need for post and core as a final restoration.
* Radiographic evidence of an apical opening width more than 2 mm with or without periapical radiolucency.
* Teeth without anatomical variations

Exclusion Criteria:• Immunocompromised patients

* Teeth with previous endodontic treatment.
* Teeth with internal or external resorption
* Radiographic evidence of root fracture.
* Lack of patient and parent cooperation.
* Presence of periodontal pocket depth more than 4 mm.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
apical closure assessed radiographically | 12 months after treatment
  radiographic evaluation of apical closure as reduction or elimination of the apical opening of the root

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry,Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
share clinical and radiograpjic outcomes with qualified researches
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication of the primary results and available for 2 years
Access Criteria: shared with qualified researchers upon reasonable request. requests should include a proposal outlining the intended use of the data
URL: https://www.tanta.edu.eg

REFERENCES:
- See also: evaluate the antimicrobial effectiveness of two irrigation medication protocols — http://www.tanta.edu.eg
- Available data/document: Study Protocol: END-7-25-3400 — http://www.tanta.edu.eg